CLINICAL TRIAL: NCT06484790
Title: An Open-Label, Dose-Escalation Phase I Clinical Study of T Cell Receptor Gene-Engineered T Cell Therapy Targeting KRAS Mutations in the Treatment of Subjects With Advanced Solid Tumor
Brief Title: T Cell Receptor Gene-Engineered T Cell Therapy Targeting KRAS Mutations in the Treatment of Subjects With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ting Deng (Other)
Collaborators: Neowise Biotechnology (Industry)
Responsible Party: Sponsor-Investigator, Ting Deng, Director, Tianjin Medical University Cancer Institute and Hospital
Organization: Tianjin Medical University Cancer Institute and Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NW-301-001
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NW-301V (Experimental): NW-301V monotherapy in patients with Solid Tumors with KRAS G12V mutation
  Interventions: Drug: NW-301V
- NW-301D (Experimental): NW-301D monotherapy in patients with Solid Tumors with KRAS G12D mutation
  Interventions: Drug: NW-301D

INTERVENTIONS:
Drug: NW-301V — TCR-T T cell targeting KRAS G12V mutation
  Arms: NW-301V
Drug: NW-301D — TCR-T T cell targeting KRAS G12D mutation
  Arms: NW-301D

SUMMARY:
An open label, two-cohort, dose-escalation clinical study to evaluate the safety, anti-tumor activity and pharmacokinetics/pharmacodynamic (PK/PD) of NW-301V and NW-301D in subjects with advanced solid tumor.

DETAILED DESCRIPTION:
Using a modified 3+3 dose escalation design, this study will enroll ~9subjects to characterize the safety and preliminary anti-tumor activity of NW-301V and NW-301D in each cohort respectively. Eligible subjects will undergo leukapheresis for autologous cell product manufacturing, and will receive a 3-day lymphodepleting regimen consisting of cyclophosphamide and fludarabine, followed by a single-dose intravenous infusion of NW-301V or NW-301D. after NW-301V or NW-301D infusion, a low dose of IL-2 will be given subcutaneously for up to 10 days. following this intervention, subjects will be monitored for safety and AE, and tumor evaluation will be performed at pre-specified timepoints per protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Age between 18-75 years
* Diagnosis of pathologically or histologically confirmed unresectable or advanced solid tumor, and have no standard treatment options available or unable to tolerate the currently available standard treatments
* HLA-A11:01positive Tumor has KRAS G12V (NW-301V cohort) or G12D (NW-301D cohort) mutation * Adequate organ function prior to apheresis and lymphodepleting chemotherapy
* ECOG performance status of 0-1
* At least one tumor lesion measurable according to RECIST 1.1 (Additional protocol-defined Inclusion criteria may apply.)

Key Exclusion Criteria:

* Received the following treatments: Cytotoxic chemotherapy within 2 weeks prior to apheresis and within 1 week prior to lymphodepletion; Treatment with antibodies (including but not limited to those with monoclonal antibodies and immune checkpoint inhibitors) or other biologic therapy within 2 weeks prior to apheresis and within 1 week prior to lymphodepletion; Immunosuppressive agents (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutic agents, mycophenolate mofetil, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti-IL-6, or anti-IL-6 receptor) within 2 weeks prior to apheresis and within 1 week prior to lymphodepletion
* History of allergic reactions to cyclophosphamide, fludarabine, or any other chemical or biological components of the drugs used in this study
* History of chronic or recurrent severe autoimmune disease, or active immune disease requiring treatment with steroids or other immunosuppressive agents within 1 year prior to enrollment* Have symptomic CNS metastases
* Have leptomeningeal disease or carcinomatous meningitis
* Have ongoing or active infection
* Active infections with HIV, HBV, HCV, or syphilis
* Breastfeeding or pregnant (Additional protocol-defined Exclusion criteria may apply.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days of single infusion
  Safety

SECONDARY OUTCOMES:
Objective response rate (ORR) | through the study completion, with average of 2 years
  complete response (CR) and partial response (PR) based on best overall response (BOR), locally assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of response (DOR) | through the study completion, with average of 2 years
  CR and PR, locally assessed using RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not provided